CLINICAL TRIAL: NCT07011927
Title: Single-center Non-inferiority Study of Extra-cochlear Electrode Placement at the Post-auricular Vagus Nerve in Cochlear Implantation
Brief Title: Extra-cochlear Electrode Placement at the Post-auricular Vagus Nerve in Cochlear Implantation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24-01768
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patients scheduled for Cochlear Implantation (Experimental): The experimental arm will enroll patients over the age of 18 undergoing cochlear implantation involving the placement of ECE1 at the approximate location of Arnold's nerve within the ear canal. In the proposed study, a modification to the surgical approach will be done to place ECE1 near Arnold's nerve, while still using a standard electrode array.
  Interventions: Device: Cochlear Implant; Device: Modified Implant Procedure

INTERVENTIONS:
Device: Cochlear Implant — Eligible Cochlear Americas devices eligible for inclusion in this study include any Cochlear Americas device that has two ground electrodes.
Device: Modified Implant Procedure — Implant procedure will be modified to place ground electrode (ECE1) near Arnold's nerve.

SUMMARY:
This study will evaluate hearing outcomes after cochlear implantation with placement of the ECE1 ground electrode near the post-auricular vagus nerve (Arnold's nerve) to assess non-inferiority with respect to placement under the temporalis muscle.

ELIGIBILITY:
Inclusion Criteria:

* will be undergoing surgery for a cochlear implant from Cochlear Americas
* is willing to participate in the study

Exclusion Criteria:

* has history of prior ear surgery, congenital ear malformation, or prior cochlear implantation in the ear to be implanted
* pregnant, planning to become pregnant, or breastfeeding patients cannot undergo the standard-of-care implantation procedures required for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-06-03 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
AzBio Sentence Recognition Test Score | Up to Year 1 post cochlear implant activation
  The AzBio Sentence Recognition Test is a clinical tool used to evaluate a person's ability to understand speech in noisy environments. The total score is the percentage of words correctly understood, ranging from 0-100%.

CONTACTS AND LOCATIONS:
Overall Officials: J. Thomas Roland, Jr., MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: mario.svirsky@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to mario.svirsky@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.